CLINICAL TRIAL: NCT05962385
Title: State Dependence of Prefrontal Transcranial Magnetic Stimulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PSYCH-2023-32060
Record Dates: First submitted 2023-07-12; First posted 2023-07-27 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Repeated measures design - across two separate sessions (one week apart, counterbalanced between participants), participants will receive transcranial magnetic stimulation (TMS) whilst engaging in either a cognitive control or a perceptual task.
Masking Description: No blinding is possible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Healthy control (Experimental): All participants receive the same procedures
  Interventions: Device: Brain state while receiving TMS

INTERVENTIONS:
Device: Brain state while receiving TMS — Brain state whilst receiving TMS - cognitive control or perceptual. Repeated measures design, so all participants receive the same procedures.

SUMMARY:
The study will examine whether the benefits of brain stimulation on mental functioning can be enhanced if an individual is actively engaging the target brain networks while receiving brain stimulation. The study includes two separate sessions and people will complete either a cognitive task or a perceptual task while receiving transcranial magnetic stimulation. The study will measure change in brain function with EEG.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65,
* healthy controls

Exclusion Criteria:

* Diagnosed psychiatric disorder
* Potential contraindications to EEG (e.g. visible scalp abrasions, non-removable hair extensions and/or hair styling that would impede proper EEG recording)
* Potential contraindication to TMS (as identified by the TMS safety screener)
* Any previous adverse reaction to TMS or MRI
* Diagnosed epilepsy or previously experienced a seizure
* Diagnosed neurological condition, such as stroke or tinnitus
* Experienced a head trauma that was diagnosed as concussion
* Current use of, or recent withdrawal from, medications that can increase the risk of seizure
* Currently pregnant
* Any metal in the head (excluding mouth)
* Any implanted medical device

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
Theta-gamma cross frequency coupling | 0-500 ms after each TMS stimulus
  A metric of brain function measured with EEG - the coupling of theta oscillation phase with gamma power. This will be measured immediately following the intervention (TMS stimulation).
Cortical excitability | 60-300 ms after each TMS stimulus
  TMS-evoked potentials will be measured with EEG to examine cortical excitability after TMS. This will be measured immediately following the intervention (TMS stimulation).

CONTACTS AND LOCATIONS:
Overall Officials: Alik Widge, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States